CLINICAL TRIAL: NCT04085367
Title: A Randomized, Double-Blind, Vehicle-Controlled, Multicenter Study to Assess the Efficacy and Safety of Methyl Aminolevulinate Hydrochloride (MAL) 16.8% Cream (CD06809-41) Versus Vehicle Cream in the Treatment of Thin and Moderately Thick, Non-hyperkeratotic, Non-pigmented Actinic Keratosis (AK) of the Face and Scalp When Using Daylight Photodynamic Therapy (DL-PDT)
Brief Title: Multicenter Study to Assess the Efficacy and Safety of Methyl Aminolevulinate Hydrochloride (MAL) 16.8% Cream (CD06809-41) Versus Vehicle Cream for Actinic Keratosis of the Face
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RD.06.SPR.112199
Record Dates: First submitted 2019-09-09; First posted 2019-09-11 (Actual); Results first posted 2022-04-01 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Actinic Keratoses
MeSH Terms: conditions — Keratosis, Actinic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MAL 16.8% Cream (Experimental): Participants received two treatment session at least 2 weeks apart. Investigator applied a thin layer of methyl aminolevulinate (MAL) hydrochloride 16.8% cream to each lesion during treatment. At 30 minutes after cream application, participants went outside in daylight for 2 hours (Daylight photodynamic therapy [DL-PDT]). After this time, the cream was removed by investigative site personnel by washing the skin with gentle skin cleanser.
  Interventions: Drug: MAL 16.8% cream
- MAL Vehicle Cream (Placebo Comparator): Participants received two treatment session at least 2 weeks apart. Investigator applied a thin layer of vehicle cream to each lesion during treatment. At 30 minutes after cream application, participants went outside in daylight for 2 hours (DL-PDT). After this time, the cream was removed by investigative site personnel by washing the skin with gentle skin cleanser.
  Interventions: Drug: MAL Vehicle Cream

INTERVENTIONS:
Drug: MAL 16.8% cream — Day light photodynamic therapy with MAL 16.8% cream
  Other Names: CD06809-41
  Arms: MAL 16.8% Cream
Drug: MAL Vehicle Cream — Day light photodynamic therapy with MAL vehicle cream
  Arms: MAL Vehicle Cream

SUMMARY:
A Randomized, Double-Blind, Vehicle-Controlled, Multicenter Study to Assess the Efficacy and Safety of Methyl aminolevulinate hydrochloride (MAL) 16.8% cream (CD06809-41) versus vehicle cream in the treatment of thin and moderately thick, non-hyperkeratotic, non-pigmented actinic keratosis of the face and scalp when using daylight photodynamic therapy (DL-PDT).

DETAILED DESCRIPTION:
This was a randomized, double-blind, vehicle-controlled, multicenter, parallel-group study in adult participants with clinically-confirmed mild to moderate AKs on the face and the balding scalp, to be conducted at approximately 60 clinical sites in the United States. Sites were selected to ensure that diverse daylight conditions represented in the study to understand the effects of latitude, elevation, and climate.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged ≥ 18 years at the Screening visit.
* Participants had at least 4, but no more than 12, clinically-confirmed thin or moderately thick, non-hyperkeratotic, non-pigmented AKs located on the face (e.g., forehead, cheek, chin), and balding scalp.
* Female Participants of non-childbearing potential.
* Participants fully understood and signed an ICF before any investigational procedure(s) are performed.

Exclusion Criteria:

* Participants with pigmented AK in the treatment areas.
* Female participants who were pregnant, nursing, or planning a pregnancy during the study.
* Participants with a clinical diagnosis of a skin disease other than AK.
* Immunocompromised participants.
* Participants with any condition that may be associated with a risk of poor protocol compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 557 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2021-03-03 (Actual); Study Completion 2021-04-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (60):
- United States (59):
  - Galderma Investigational Site (Site 8768), Tucson, Arizona
  - Galderma Investigational Site (Site 8447), Fort Smith, Arkansas
  - Galderma Investigational Site (Site 8577), Encinitas, California
  - Galderma Investigational Site (Site 8636), Fountain Valley, California
  - Galderma Investigational Site (Site 8224), Fremont, California
  - Galderma Investigational Site (Site 8114), Fresno, California
  - Galderma Investigational Site (Site 8758), San Diego, California
  - Galderma Investigational Site (Site 8608), Santa Monica, California
  - Galderma Investigational Site (Site 8778), Denver, Colorado
  - Galderma Investigational Site (Site 8440), Greenwood Village, Colorado
  - Galderma Investigational Site (Site 8479), Bradenton, Florida
  - Galderma Investigational Site (Site 8770), Lehigh Acres, Florida
  - Galderma Investigational Site (Site 8656), Miami, Florida
  - Galderma Investigational Site (Site 8765), North Miami Beach, Florida
  - Galderma Investigation Site (Site 8769), Palm Springs, Florida
  - Galderma Investigational Site (Site 8734), Pembroke Pines, Florida
  - Galderma Investigational Site (Site 8529), Sanford, Florida
  - Galderma Investigational Site (Site 8126), West Palm Beach, Florida
  - Galderma Investigational Site (Site 8683), Atlanta, Georgia
  - Galderma Investigational Site (Site 8860), Atlanta, Georgia
  - Galderma Investigational Site (Site 8667), Columbus, Georgia
  - Galderma Investigational Site (Site 8755), Boise, Idaho
  - Galderma Investigational Site (Site 8838), Darien, Illinois
  - Galderma Investigational Site (Site 8724), Louisville, Kentucky
  - Galderma Investigational Site (Site 8208), Beverly, Massachusetts
  - Galderma Investigational Site (Site 8574), Clarkston, Michigan
  - Galderma Investigation Site (Site 8757), Saint Joseph, Michigan
  - Galderma Investigational Site (Site 8762), Edina, Minnesota
  - Galderma Investigational Site (Site 8140), New Brighton, Minnesota
  - Galderma Investigational Site (Site 8219), St Louis, Missouri
  - Galderma Investigational Site (Site 8869), St Louis, Missouri
  - Galderma Investigational Site (Site 8048), Omaha, Nebraska
  - Galderma Investigational Site (Site 8420), Portsmouth, New Hampshire
  - Galderma Investigational Site (Site 8759), Albuquerque, New Mexico
  - Galderma Investigational Site (Site 8242), Brooklyn, New York
  - Galderma Investigational Site (Site 8733), New York, New York
  - Galderma Investigational Site (Site 8279), New York, New York
  - Galderma Investigational Site (Site 8566), Charlotte, North Carolina
  - Galderma Investigational Site (Site 8726), Wilmington, North Carolina
  - Galderma Investigational Site (Site 8595), Dublin, Ohio
  - Galderma Investiational Site (Site 8212), Portland, Oregon
  - Galderma Investigational Site (Site 8255), Philadelphia, Pennsylvania
  - Galderma Investigational Site (Site 8721), Pittsburgh, Pennsylvania
  - Galderma Investigational Site (Site 8754), Sugarloaf, Pennsylvania
  - Galderma Investigational Site (Site 8777), Charleston, South Carolina
  - Galderma Investigational Site (Site 8207), Nashville, Tennessee
  - Galderma Investigational Site (Site 8076), Austin, Texas
  - Galderma Investigational Site (Site 8139), College Station, Texas
  - Galderma Investigational Site (Site 8664), Frisco, Texas
  - Galderma Investigational Site (Site # 8576), Houston, Texas
  - Galderma Investigational Site (Site 8546), Pflugerville, Texas
  - Galderma Investigational Site (Site 8672), Salt Lake City, Utah
  - Galderma Investigational Site (Site 8776), St. George, Utah
  - Galderma Investigational Site (Site 8761), West Jordan, Utah
  - Galderma Investigational Site (Site 8057), Lynchburg, Virginia
  - Galderma Investigational Site (Site 8779), Burien, Washington
  - Galderma Investigational Site (Site 8039), Spokane, Washington
  - Galderma Investigational Site (Site 8760), Spokane, Washington
  - Galderma Investigational Site (Site 8725), Morgantown, West Virginia
- Galderma Investigational Site (Site 8231), Aibonito, Puerto Rico

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 557 participants were randomized in 2:1 ratio in two treatment group, MAL 16.8% cream and vehicle cream in study centers in the United States with diverse latitude, altitude, and climate characteristics.
Period: Overall Study
Arm/Group | MAL 16.8% Cream | MAL Vehicle Cream
Started | 364 | 193
Completed | 344 | 185
Not Completed | 20 | 8
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 13 | 4
Not completed — Lost to Follow-up | 3 | 1
Not completed — Other unspecified | 2 | 1
Not completed — Status Unknown | 1 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) analysis population included all participants randomized in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | MAL 16.8% Cream | MAL Vehicle Cream | Total
Number analyzed (Participants) | 364 | 193 | 557
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.2 (8.75) | 68.9 (9.00) | 69.1 (8.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 61 | 159
  Male | 266 | 132 | 398
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 15 | 48
  Not Hispanic or Latino | 327 | 177 | 504
  Unknown or Not Reported | 4 | 1 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 0 | 2
  White | 359 | 192 | 551
  More than one race | 1 | 1 | 2
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Complete Response at Week 12
Description: Complete response was defined as clearance of all AK lesion treated, at week 12 after the last Daylight photodynamic therapy (DL-PDT).
Time Frame: Week 12
Population: ITT analysis population included all participants randomized in the study.
Measure: Number; unit: percentage of participants
Groups:
- MAL 16.8% Cream: Participants received two treatment session at least 2 weeks apart. Investigator applied a thin layer of methyl aminolevulinate (MAL) hydrochloride 16.8% cream to each lesion. At 30 minutes after cream application, participants went outside in daylight for 2 hours (Daylight photodynamic therapy [DL-PDT]). After this time, the cream was removed by investigative site personnel by washing the skin with gentle skin cleanser.
- MAL Vehicle Cream: Participants received two treatment session at least 2 weeks apart. Investigator applied a thin layer of vehicle cream to each lesion. At 30 minutes after cream application, participants went outside in daylight for 2 hours (DL-PDT). After this time, the cream was removed by investigative site personnel by washing the skin with gentle skin cleanser.
Arm/Group | MAL 16.8% Cream | MAL Vehicle Cream
Number analyzed (Participants) | 364 | 193
percentage of participants | 25.3 | 23.0

2. Secondary Outcome: Percent Change From Baseline in Lesion Complete Response at Week 12
Description: Lesion complete response was defined as percent reduction from baseline in the number of cleared treated lesions, at 12 weeks after the last DL-PDT treatment. This outcome measure was analyzed as an intra-individual comparison between MAL cream and Vehicle cream.
Time Frame: Baseline, Week 12
Population: ITT analysis population included all participants randomized in the study.
Measure: Mean (Standard Error); unit: percent change
Arm/Group | MAL 16.8% Cream | MAL Vehicle Cream
Number analyzed (Participants) | 364 | 193
percent change | -61.1 (1.79) | -49.4 (2.45)

3. Secondary Outcome: Percentage of Participants With Partial Response at Week 12
Description: Participants achieving partial response was defined as participants with 75% or greater reduction from baseline in the number of cleared treated lesions, at 12 weeks after the last DL-PDT treatment, comparing MAL cream with vehicle cream.
Time Frame: Week 12
Population: ITT analysis population included all participants randomized in the study.
Measure: Number; unit: percentage of participants
Arm/Group | MAL 16.8% Cream | MAL Vehicle Cream
Number analyzed (Participants) | 364 | 193
percentage of participants | 48.2 | 35.1

ADVERSE EVENTS:
Time Frame: Baseline up to Week 14
Description: Safety population consisted of all randomized participants who received at least 1 application of study drug.
Groups:
- MAL 16.8% Cream: Participants received two treatment session at least 2 weeks apart. Investigator was to apply a thin layer of methyl aminolevulinate (MAL) hydrochloride 16.8% cream to each lesion during treatment. At 30 minutes after cream application, participants were to go outside in daylight for 2 hours. After this time, the cream was to be removed by investigative site personnel by washing the skin with gentle skin cleanser.
- MAL Vehicle Cream: Participants received two treatment session at least 2 weeks apart. Investigator was to apply a thin layer of vehicle cream to each lesion during treatment. At 30 minutes after cream application, participants were to go outside in daylight for 2 hours. After this time, the cream was to be removed by investigative site personnel by washing the skin with gentle skin cleanser.
Arm/Group | MAL 16.8% Cream | MAL Vehicle Cream
All-Cause Mortality (participants affected / at risk) | 0/364 | 0/193
Serious Adverse Events (participants affected / at risk) | 5/364 | 1/193
Other Adverse Events (participants affected / at risk) | 89/364 | 41/193
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MAL 16.8% Cream (N=364) | MAL Vehicle Cream (N=193)
Back injury (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Streptococcal endocarditis (Infections and infestations) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MAL 16.8% Cream (N=364) | MAL Vehicle Cream (N=193)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 62 | 30
Skin lesion (Skin and subcutaneous tissue disorders) | 4 | 2
Application site pain (General disorders) | 11 | 2
Application site erythema (General disorders) | 12 | 0
Application site dermatitis (General disorders) | 7 | 1
Application site pruritus (General disorders) | 5 | 3
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 7 | 3
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2020-07-12): https://cdn.clinicaltrials.gov/large-docs/67/NCT04085367/Prot_000.pdf
  • Statistical Analysis Plan (2021-04-06): https://cdn.clinicaltrials.gov/large-docs/67/NCT04085367/SAP_001.pdf